CLINICAL TRIAL: NCT03850119
Title: Nanofat on Wound Healing and Scar Formation: a Randomized, Split-scar, Double Blind Trial
Brief Title: Nanofat on Wound Healing and Scar Formation
Acronym: NFWHSF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Moustapha Hamdi, Head of department Plastic and Reconstructive surgery, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-044
Record Dates: First submitted 2019-02-18; First posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Scars; Delayed Wound Healing; Hypertrophic Scar; Post Inflammatory Hyperpigmentation; Donor Site Complication
Keywords: adipose derived stem cells; stromal vascular fraction; wound healing; scar formation; donor site morbidity; nanofat
MeSH Terms: conditions — Cicatrix; Cicatrix, Hypertrophic; Hyperpigmentation

STUDY DESIGN:
Intervention Model Description: monocentric randomized controlled double-blinded prospective interventional study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patient, investigator, outcome assessor will be blinded for which side of the scar was treated and which was a control. Only the surgeon, who will not be involved in the assessment, will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intradermal Nanofat (Experimental): This side of the scar received intradermal injection of nanofat during the closure of the donor site.
  Interventions: Procedure: Nanofat injection
- Control (No Intervention): This side of the scar received no injection.

INTERVENTIONS:
Procedure: Nanofat injection — Lipoaspirate, harvested during the surgery, is centrifuged for 1 minute at 2000 rpm to discard infiltration fluid. The residual fat is passed back and forth between two 10cc syringes interlocked with Tulip connecting pieces (2.4, 1.4 and 1.2 diameter, each 10 passes for a total of 30 passes). This is injected intradermally before the intradermal sutures are placed. The donor site is always entirely sutured (both sides) by the same person.
  Arms: Intradermal Nanofat

SUMMARY:
This study will evaluate the effectiveness and safety of intradermal injection of Nanofat on wound healing and scar formation.

DETAILED DESCRIPTION:
In this monocentric, randomized, controlled, double-blinded prospective interventional study, twenty patients will be included. Each patient will be his/her own control.

Patients undergoing DIEPflap breast reconstruction will be included in this study. During the surgery, the abdominal incision will be divided in two equal sides with the umbilicus as midline reference. The sides will be randomized in a treatment side and control side. The treatment side will receive intradermal nanofat injections after the subcutaneous and right before the intradermal sutures.

The patient and investigators will be blinded for the treatment protocol. The effects on wound healing, adverse events, scar formation and pigmentation will be evaluated up to one year after the surgery.

ELIGIBILITY:
Inclusion Criteria:

- scheduled for DIEP-flap breast reconstruction surgery at our department

Exclusion Criteria:

* smokers
* use of cortisone or other immunsuppressants
* diabetes mellitus type 1 or 2
* age
* connective tissue disease

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome of the abdominal scar by the use of Patient and Observer Scar Assessment Scale | one year
  The abdominal scar will be evaluated clinically by the patient and observer scar assessment scale, starting from one month after the surgery
Clinical assessment of the time to healing of the abdominal wound | one month
  The time for the abdominal wound to heal will be registered. Wound healing is considered a closed and non-dehiscent wound witout signs of inflammation or infection.
Evaluation of histological parameters on tissue biopsy from both sides of the abdominal scar. | six months
  Evaluation of the histological differences of the treatment arm vs. control, by evaluating scar properties on tissue biopsy. Scar thickness, collagen arrangement and angiogenesis will be evaluated.
Pigmentation Index of the two sides of the scar, measured with a Mexameter | one year
  Evaluation of the Pigmentation Index difference in the treatment arm vs. control arm will be measured by the use of a mexameter, starting from one month after the procedure (after wound healing is complete).
Patient satisfaction of abdominal scar appearance measured by a Visual Analog Scale | one year
  Evaluation of patient satisfaction over the entire course of the study by filling in a Visual Analog Scale, with 1 being very unsatisfied and 10 being very satisfied.
Rate of adverse events | One year
  Registration of the rate of adverse events appearing at the abdominal wound/abdominal scar

CONTACTS AND LOCATIONS:
Overall Officials: Moustapha Hamdi, MD,PhD, Principal Investigator — Universitair Ziekenhuis Brussel

IPD SHARING:
Plan to Share IPD: No